CLINICAL TRIAL: NCT00613756
Title: Post Marketing Surveillance of BI-Sifrol® (Pramipexole). Special Survey on Patients With Parkinson's Disease and Renal Dysfunction
Brief Title: Special Survey on PD Patients With Renal Dysfunction
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 248.548
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The survey is conducted to collect safety and effectiveness information targeting patients who have both Parkinson's disease and renal dysfunction treated with Pramipexole in the daily clinical settings in Japan.

ELIGIBILITY:
Inclusion Criteria:

Patients with Parkinson's disease who have renal dysfunction with pretreatment creatinine clearance =<70mL/min or whose renal dysfunction was determined by the physician

Exclusion Criteria:

None

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with idiopathic PD with renal dysfunction from Primary Care setting.
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2004-02; Primary Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | up to 12 weeks
Incidence of adverse drug reactions (ADRs | up to 12 weeks
Incidence of serious adverse events (SAEs) | up to 12 weeks

SECONDARY OUTCOMES:
Modified Hoehn & Yahr rating scale | change from baseline to week 12
Unified Parkinson's Disease Rating Scale (UPDRS) part III total score | change from baseline to week 12
Physician's overall judgement by medical interview into 4 grades (5 categories) | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (97):
- Japan (97):
  - Boehringer Ingelheim Investigational Site, Asahikawa
  - Boehringer Ingelheim Investigational Site, Azumino
  - Boehringer Ingelheim Investigational Site, Chūō
  - Boehringer Ingelheim Investigational Site, Fuji
  - Boehringer Ingelheim Investigational Site, Fujinomiya
  - Boehringer Ingelheim Investigational Site, Fujisaki
  - Boehringer Ingelheim Investigational Site, Fukaya
  - Boehringer Ingelheim Investigational Site, Fukui
  - Boehringer Ingelheim Investigational Site, Fukuoka
  - Boehringer Ingelheim Investigational Site, Gifu
  - Boehringer Ingelheim Investigational Site, Hachiōji
  - Boehringer Ingelheim Investigational Site, Hamamatsu
  - Boehringer Ingelheim Investigational Site, Himeji
  - Boehringer Ingelheim Investigational Site, Hiroshima
  - Boehringer Ingelheim Investigational Site, Ichinoseki
  - Boehringer Ingelheim Investigational Site, Iga
  - Boehringer Ingelheim Investigational Site, Iida
  - Boehringer Ingelheim Investigational Site, Iijima
  - Boehringer Ingelheim Investigational Site, Ina
  - Boehringer Ingelheim Investigational Site, Inazawa
  - Boehringer Ingelheim Investigational Site, Isehara
  - Boehringer Ingelheim Investigational Site, Isesaki
  - Boehringer Ingelheim Investigational Site, Iwamizawa
  - Boehringer Ingelheim Investigational Site, Kagoshima
  - Boehringer Ingelheim Investigational Site, Kajiki
  - Boehringer Ingelheim Investigational Site, Kanoya
  - Boehringer Ingelheim Investigational Site, Kashiwazaki
  - Boehringer Ingelheim Investigational Site, Kawagoe
  - Boehringer Ingelheim Investigational Site, Kawasaki
  - Boehringer Ingelheim Investigational Site, Koga
  - Boehringer Ingelheim Investigational Site, Komae
  - Boehringer Ingelheim Investigational Site, Koshigaya
  - Boehringer Ingelheim Investigational Site, Kōriyama
  - Boehringer Ingelheim Investigational Site, Kurashiki
  - Boehringer Ingelheim Investigational Site, Kyoto
  - Boehringer Ingelheim Investigational Site, Maebashi
  - Boehringer Ingelheim Investigational Site, Marugame
  - Boehringer Ingelheim Investigational Site, Matsudo
  - Boehringer Ingelheim Investigational Site, Matsumoto
  - Boehringer Ingelheim Investigational Site, Miki
  - Boehringer Ingelheim Investigational Site, Mito
  - Boehringer Ingelheim Investigational Site, Miyazaki
  - Boehringer Ingelheim Investigational Site, Miyoshi
  - Boehringer Ingelheim Investigational Site, Mooka
  - Boehringer Ingelheim Investigational Site, Morioka
  - Boehringer Ingelheim Investigational Site, Morohongō
  - Boehringer Ingelheim Investigational Site, Nagahama
  - Boehringer Ingelheim Investigational Site, Nagakute
  - Boehringer Ingelheim Investigational Site, Nagasaki
  - Boehringer Ingelheim Investigational Site, Nagoya
  - Boehringer Ingelheim Investigational Site, Nanao
  - Boehringer Ingelheim Investigational Site, Nangōku
  - Boehringer Ingelheim Investigational Site, Narita
  - Boehringer Ingelheim Investigational Site, Nishinomiya
  - Boehringer Ingelheim Investigational Site, Okayama
  - Boehringer Ingelheim Investigational Site, Okinawa
  - Boehringer Ingelheim Investigational Site, Osaka
  - Boehringer Ingelheim Investigational Site, Ōgaki
  - Boehringer Ingelheim Investigational Site, Ōita
  - Boehringer Ingelheim Investigational Site, Ōkawa
  - Boehringer Ingelheim Investigational Site, Ōnojō
  - Boehringer Ingelheim Investigational Site, Ōshū
  - Boehringer Ingelheim Investigational Site, Sado
  - Boehringer Ingelheim Investigational Site, Sagamihara
  - Boehringer Ingelheim Investigational Site, Saitama
  - Boehringer Ingelheim Investigational Site, Sanjō
  - Boehringer Ingelheim Investigational Site, Sapporo
  - Boehringer Ingelheim Investigational Site, Sekigahara
  - Boehringer Ingelheim Investigational Site, Shimotsuke
  - Boehringer Ingelheim Investigational Site, Shingū
  - Boehringer Ingelheim Investigational Site, Shūnan
  - Boehringer Ingelheim Investigational Site, Suita
  - Boehringer Ingelheim Investigational Site, Takasago
  - Boehringer Ingelheim Investigational Site, Takatsuki
  - Boehringer Ingelheim Investigational Site, Togitsu
  - Boehringer Ingelheim Investigational Site, Tokyo Adachi-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Bunkyo-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Chiyoda-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Itabashi-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Meguro-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Ota-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Setagaya-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Shibuya-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Shinjuku-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Suginami-ku
  - Boehringer Ingelheim Investigational Site, Toride
  - Boehringer Ingelheim Investigational Site, Toyoake
  - Boehringer Ingelheim Investigational Site, Tsukuba
  - Boehringer Ingelheim Investigational Site, Uki
  - Boehringer Ingelheim Investigational Site, Wakayama
  - Boehringer Ingelheim Investigational Site, Yamagata
  - Boehringer Ingelheim Investigational Site, Yamaguchi
  - Boehringer Ingelheim Investigational Site, Yokohama
  - Boehringer Ingelheim Investigational Site, Yokosuka
  - Boehringer Ingelheim Investigational Site, Yonago
  - Boehringer Ingelheim Investigational Site, Yoshinogawa
  - Boehringer Ingelheim Investigational Site, Yufu